CLINICAL TRIAL: NCT02662998
Title: Validation of uHear™ as a Screening Tool to Detect Hearing Impairment in Older Cancer Patients Within a Comprehensive Geriatric Assessment - BIS
Acronym: UHEAR-BIS
Status: Completed | Type: Observational
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Medical Oncologist, General Hospital Groeninge
Other Study IDs: AZGS2015133
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Older Cancer Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of this study is to validate uHear™, an iOS-based tool, as a screening tool to detect significant hearing impairment as part of a comprehensive geriatric assessment in patients aged 70 years and older. The pass or fail screening cut-off is defined as having two or more consecutive hearing grades starting from the moderate-severe threshold zone ranging from 0.5 - 2.0 kHz.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have reached the age of 70 or more at enrolment
* Histologically confirmed diagnosis of solid cancer or hematologic malignancy. All stages of cancer are eligible
* Patients should be fluent in Dutch or French
* Patients must receive their primary oncology care in the participating hospital
* Patients should be cognitively capable of performing the audiology assessment
* Patients should be scheduled to receive a CGA
* Patients should have signed informed consent

Exclusion Criteria:

* Patients who do not match the above inclusion criteria
* Patients presenting with clinically diagnosed Meniere's disease, retrocochlear hearing loss, autoimmune inner ear disease, fluctuating hearing loss or a history of sudden sensory neural hearing loss
* Patients who already have a hearing aid or a previously diagnosed hearing loss

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This trial will recruit older patients with a minimum age of 70 years old who have been diagnosed with a solid tumour or hematologic malignancy, who are eligible for an oncogeriatric evaluation.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Validation of uHear™ with its new scoring method as a screening tool to detect hearing loss in older cancer patients | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Groeninge, Cancer Center, Kortrijk, Belgium

REFERENCES:
- [Result] Lycke M, Debruyne PR, Lefebvre T, Martens E, Ketelaars L, Pottel H, Van Eygen K, Derijcke S, Werbrouck P, Vergauwe P, Stellamans K, Clarysse P, Dhooge I, Schofield P, Boterberg T. The use of uHear to screen for hearing loss in older patients with cancer as part of a comprehensive geriatric assessment. Acta Clin Belg. 2018 Apr;73(2):132-138. doi: 10.1080/17843286.2017.1392070. Epub 2017 Oct 24. PMID 29063810